CLINICAL TRIAL: NCT04068168
Title: Open Label, Multicenter, Real World Practice of Durvalumab (Imfinzi PMS)
Acronym: Imfinzi PMS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4194R00004
Record Dates: First submitted 2019-08-07; First posted 2019-08-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer, Biliary Tract Cancer
MeSH Terms: conditions — Lung Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The objectives of this study are to assess safety and efficacy of Imfinzi (durvalumab) in a real world setting in patients treated with Imfinzi under the approved indication in Korea.

DETAILED DESCRIPTION:
Primary objective : To assess safety of Imfinzi for patients treated with Imfinzi under the approved indication in Korea

Outcome Measure:

* Safety (adverse event (AE), serious adverse events (SAE), adverse drug reaction (ADR), serious adverse drug reaction (SADR), adverse events of special interest (AESI), adverse events leading to discontinuation (DAE), and adverse events leading to deaths (fatal AE))
* Dose interruptions
* Duration of treatment
* Reason for treatment discontinuation Secondary objective: To assess efficacy of Imfinzi for patients treated with Imfinzi under the approved indication in Korea

Outcome Measure:

* Progression free survival (PFS)
* Objective response rate (ORR)
* Duration of response (DoR)

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Imfinzi treatment according to the approved label
* Provision of signed and dated written informed consent by the patient or legally acceptable representative

Exclusion Criteria:

* Current participation in any interventional trial
* Other off-label indications according to the approved label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Imfinzi treatment according to the approved label
Sampling Method: Non-Probability Sample
Enrollment: 712 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Safety (AE, SAE, ADR, SADR, AESI, DAE, fatal AE) | for up to 1 year after the first dose of Imfinzi
  safety outcome
Dose interruptions | for up to 1 year after the first dose of Imfinzi
  Safety outcome
Duration of treatment | for up to 1 year after the first dose of Imfinzi
  Safety outcome

SECONDARY OUTCOMES:
Progression free survival (PFS) | for up to 1 year after the first dose of Imfinzi
  efficacy outcome
Objective response rate (ORR) | for up to 1 year after the first dose of Imfinzi
  efficacy outcome
Duration of response (DoR) | for up to 1 year after the first dose of Imfinzi
  efficacy outcome

CONTACTS AND LOCATIONS:
Locations (24):
- South Korea (24):
  - Research Site, Anyang-si, South Korea
  - Research Site, Bucheon-si, South Korea
  - Research Site, Busan, South Korea
  - Research Site, Changwon, South Korea
  - Research Site, Changwon-si, South Korea
  - Research Site, Cheonan, South Korea
  - Research Site, Chuncheon, South Korea
  - Research Site, Daegu, South Korea
  - Research Site, Daejeon, South Korea
  - Research Site, Goyang-si, South Korea
  - Research Site, Gwangju, South Korea
  - Research Site, Hwasun-gun, South Korea
  - Research Site, Iksan-si, South Korea
  - Research Site, Incheon, South Korea
  - Research Site, Jeju-do, South Korea
  - Research Site, Jeonju, South Korea
  - Research Site, Pohang-si, South Korea
  - Research Site, Seongnam-si, South Korea
  - Research Site, Seoul, South Korea
  - Research Site, Suwon, South Korea
  - Research Site, Uijeongbu-si, South Korea
  - Research Site, Wŏnju, South Korea
  - Research Site, Yangsan, South Korea
  - Research Site, Yongin-si, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194R00004&attachmentIdentifier=95177cc7-3dc5-4f80-83f5-a1141ed6686f&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=